CLINICAL TRIAL: NCT07314632
Title: Prospective Study on the Incidence of Recurrence in Laser Treatment of Pilonidal Cysts
Brief Title: Prospective Study in Laser Treatment of Pilonidal Cysts
Acronym: LASPRO
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CH25_0098; 2025-A02356-43 (Other: national registration number)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pilonidal Sinus
Keywords: Pilonidal sinus; laser; risk factors; Recurrence rates
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients requiring laser surgery for pilonidal sinus: pilonidal sinus of any type (including recurrence after radical cure or laser treatment)

SUMMARY:
The goal of this observational study is to evaluate the recurrence rate after laser treatment of pilonidal sinus within two years of the procedure in adult patients who require this procedure to treat their pilonidal sinus.

The main question it aims to answer is:

• Is there a clinical recurrence (presence of a fistula in the intergluteal cleft) 2 years after laser treatment of pilonidal sinus? Participants who undergo surgery as part of their regular medical care will answer survey questions about recurrence at 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring laser surgery for pilonidal sinus, of any type (including recurrence after radical cure or laser treatment)
* Patient able to understand the protocol and having given written informed consent to participate in the study,
* Patient affiliated to the social security system or entitled to it.

Exclusion Criteria:

* Patient participating in another interventional clinical research protocol involving a drug or clinical investigation of a medical device
* Patient already included in a research study
* Patient under guardianship, conservatorship, or deprived of liberty
* Patient under an activated future protection mandate
* Patient under family authorization
* Patient under judicial protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in two centers that regularly perform laser treatment for pilonidal cysts.
  Recruitment will be conducted prospectively upon the patients' arrival at the digestive surgery department.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2030-06-12 (Estimated); Study Completion 2030-06-12 (Estimated)

PRIMARY OUTCOMES:
Clinical recurrence | 2 years post-operatively
  2-year recurrence rate after laser sinusectomy (presence of openings in the intergluteal cleft)

CONTACTS AND LOCATIONS:
Overall Officials: Tristan GREILSAMER, PH, Principal Investigator — Centre Hospitalier Departemental Vendée
Locations (2):
- France (2):
  - Clinique des Cèdres, Cornebarrieu
  - CHD Vendée, La Roche-sur-Yon

IPD SHARING:
Plan to Share IPD: No